CLINICAL TRIAL: NCT05928780
Title: A Molecular Pathway-based Umbrella Trial for First-line Precision Therapy With TROP2 in Patients With Locally Advanced or Metastatic TNBC (Future-Trop2 Study)
Brief Title: An Umbrella Trial Based on Molecular Pathway for Patients With Metastatic TNBC in First-line Treatment (FUTURE-Trop2)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Future-Trop2
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LAR (Experimental): Coelomofacial androgen receptor
  Interventions: Drug: A1:SG with SHR3680; Drug: A2:SG
- IM (Experimental): Immunoregulatory type
  Interventions: Drug: B1:SG with SHR1210; Drug: B2:SG
- BLIS (Experimental): Basal type and immunosuppressive type
  Interventions: Drug: C1:SG with SHR3162; Drug: C2:SG
- MES (Experimental): Interstitial type
  Interventions: Drug: D1:SG with VEGFRI; Drug: D2:SG

INTERVENTIONS:
Drug: A1:SG with SHR3680 — SG 10mg/kg d1, 8；SHR3680 240mg qd，3 weeks is a cycle
  Arms: LAR
Drug: A2:SG — SG 10mg/kg d1, 8
  Arms: LAR
Drug: B1:SG with SHR1210 — SG 10mg/kg， d1, 8；SHR1210 200mg，d1，q3w；
  Arms: IM
Drug: B2:SG — SG 10mg/kg， d1, 8
  Arms: IM
Drug: C1:SG with SHR3162 — SG 10mg/kg d1, 8；SHR3162，150mg，QD ，3 weeks is a cycle
  Other Names: Phase Ib dose ramp
  Arms: BLIS
Drug: C2:SG — SG 10mg/kg d1, 8
  Arms: BLIS
Drug: D1:SG with VEGFRI — SG 10mg/kg，d1, 8；BP102 15mg/kg，d1，3 weeks is a cycle
  Other Names: Phase Ib dose ramp
  Arms: MES
Drug: D2:SG — SG 10mg/kg d1, 8
  Arms: MES

SUMMARY:
To explore the efficacy and safety of TROP2 in the treatment of ABC

DETAILED DESCRIPTION:
To explore the efficacy and safety of advanced first-line TROP2 precision therapy in patients with locally advanced or metastatic triple-negative breast cancer based on molecular subtypes

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old and ≤70 years old.
* ECOG body status level 0 ~ 1.
* The expected survival is not less than 3 months.
* Breast cancer patients with histologically proven invasive triple-negative breast cancer (specifically defined as estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER-2) who are all negative by pathological tests. Specifically: ER negative: IHC<1%, PR negative: IHC<1%, HER2 negative: IHC-/+ or IHC++ but FISH/CISH negative. All specimens should be verified by the pathology department of the research center, and the molecular typing of relapses and metastases should be re-checked.
* Tumor stage: recurrent or metastatic breast cancer; Patients with local recurrence need to be confirmed by the investigator that radical surgical resection is not possible.
* Stage II: patients who have not used paclitaxel or have used paclitaxel in adjuvant/neoadjuvant therapy, but the interval from the end of treatment to relapse is greater than 6 months; No systemic anti-tumor therapy (chemotherapy, targeted therapy, etc.) has been received in the advanced stage.
* Stage I: The advanced stage has received ≥1 line systemic anti-tumor therapy (chemotherapy, targeted therapy, etc.).
* Have at least one measurable lesion or unmeasurable lesion according to RECIST version 1.1 (measurable lesion ≥20mm conventional CT scan and ≥10mm spiral CT scan, measurable lesion not receiving radiotherapy).
* The functions of the main organs are basically normal.
* Have not received radiotherapy, endocrine therapy, molecular targeted therapy, or surgery (except for procedures unrelated to antitumor therapy such as central venous catheterization) within 3 weeks prior to the start of the study, and have recovered from acute toxic effects of previous treatment (if surgery is available, the wound has fully healed).
* No peripheral neuropathy or grade I peripheral neurotoxicity.
* Fertile female subjects are required to use a medically approved contraceptive during study treatment and for at least 3 months after the last use of the study drug; The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Stage II: patients with adjuvant/neoadjuvant use of paclitaxel but the interval from the end of taxol treatment to recurrence and metastasis is less than 6 months, or have received systemic anti-tumor therapy (chemotherapy, targeted therapy, etc.) in the late stage;
* Stage I: no systemic anti-tumor therapy (chemotherapy, targeted therapy, etc.) has been received in the advanced stage;
* Patients with known central nervous system metastasis or history of central nervous system metastasis prior to screening. For patients with clinically suspected central nervous system metastasis, enhanced CT or enhanced Magnetic Resonance Imaging (MRI) must be performed within 28 days before the first dose to rule out central nervous system metastasis.
* A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
* Persistent grade ≥1 adverse events due to previous treatment. The exception to this is hair loss or something the researchers believe should not be ruled out. Such cases should be clearly documented in the investigator's notes;
* Major surgery was performed within 3 weeks of the first course of trial treatment (except for minor outpatient surgery, such as placement of vascular access);
* Pregnant or lactating patients;
* Other malignancies within the previous 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or skin squamous cell carcinoma.
* Inability to swallow, chronic diarrhea and intestinal obstruction, there are multiple factors that affect drug use and absorption;
* There is a third space effusion that cannot be controlled by drainage or other methods (such as excessive pleural fluid and ascites);
* Participated in clinical trials of other antitumor drugs within 4 weeks before taking the study drug for the first time;
* long-term unhealed wounds or incomplete healing fractures;
* Patients with known HBV or HCV infection active phase or hepatitis B DNA≥500, or chronic phase with abnormal liver function;
* Allergic physique, or known allergic history of the drug components of this program; Or allergic to other monoclonal antibodies;
* Malignant tumors within the past five years (except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 125 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
PFS | max 6 months
  time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
OS | max 6 months
  Overall survival
ORR | max 6 months
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
DOR | max 6 months
  Duration of Overall Response.The date of the first assessed PR/CR (according to RECIST 1.1) to the date of the first assessed tumor progression (according to RECIST 1.1) or death from any cause.